CLINICAL TRIAL: NCT06655181
Title: Investigation of the Effectiveness of Respiratory Muscle Training in Children With Kidney Transplantation
Brief Title: Evaluating the Effectiveness of Respiratory Muscle Training in Pediatric Kidney Transplant Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Meltem Kaya, Assistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AtlasUmkaya03
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease(CKD); Pediatric ALL; Pediatric Kidney Transplantation; Respiratory Muscle Training
Keywords: Pediatric kidney transplantation; respiratory muscle training
MeSH Terms: conditions — Renal Insufficiency, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in the experimental group will be taught a home-based chest physiotherapy program (breathing exercises, teaching relaxation positions, cough training, respiratory control, respiratory control, physical activity recommendation) to be applied for 30 minutes a day, 5 days a week for 8 weeks. In addition to this program, the participants in the experimental group will be given inspiratory and expiratory combined respiratory muscle training at 30% of MEP and MIP values for 8 weeks, 2 times a day for 20 minutes each, at least 5 days a week. The resistance setting of the participants in the experimental group will be adjusted to be calculated by measuring MIP-MEP again.
  Interventions: Device: Respiratory Muscle Training
- Control Group (Sham Comparator): Participants in the control group will be taught a home-based chest physiotherapy program (breathing exercises, teaching relaxation positions, cough training, respiratory control, respiratory control, physical activity recommendation) to be applied for 30 minutes a day, 5 days a week for 8 weeks. Patients in the control group will receive sham combined respiratory muscle training at the lowest constant load, twice a day for 20 minutes each, at least 5 days a week for a total of 8 weeks.
  Interventions: Device: Respiratory Muscle Training

INTERVENTIONS:
Device: Respiratory Muscle Training — Expiratory muscle training will be performed with POWERbreathe EX1 Medic (POWERbreathe®) device and inspiratory muscle training will be performed with POWERbreathe Medic Classic device.

SUMMARY:
Chronic kidney disease is defined as kidney damage lasting three months or longer and irreversible loss of renal function (glomerular, tubular and endocrine) or a glomerular filtration rate of less than 60 ml/min /1.73 m2 . Among the five stages of chronic kidney disease, the last and most severe stage is end-stage chronic kidney disease, which requires kidney transplantation. Many organs and systems are affected after kidney transplantation. Anemia, cardiovascular complications, secondary hyperparathyroidism, accumulation of uremic toxins, electrolyte disturbances, uremic myopathy, vitamin D deficiency, malnutrition, inflammation, atherosclerosis syndrome, and respiratory dysfunction and respiratory muscle weakness caused by oxidative stress leading to loss of muscle tissue are the most common changes seen in the pulmonary system. Children undergoing transplantation are at higher risk for cardiovascular diseases, usually associated with hypertension and dyslipidemia, which are already present in the chronic kidney disease stage and persist after transplantation. Significantly reduced muscle strength and physical activity in pediatric kidney transplant recipients is also frequently reported in the literature. Decreased exercise capacity, muscle strength and physical activity increase the risk of pulmonary and cardiovascular diseases. As chronic kidney disease progresses, pulmonary complications such as restrictive pulmonary dysfunction, respiratory muscle myopathy and decreased respiratory muscle strength are associated with disease severity. To improve respiratory muscle strength, respiratory muscle training is recommended for people with chronic kidney disease. The literature has so far demonstrated positive effects of inspiratory muscle training on respiratory muscle strength, diaphragm thickness and mobility, lung volumes, functional capacity and quality of life in many other patient populations, including lung and heart disease, cardiac surgery, thoracic surgery, multiple sclerosis and stroke. Although recent studies have found evidence of systemic changes after transplantation in both adults and children, there is little evidence of the efficacy of respiratory muscle training, especially in pediatric patients. In the light of all this information, the aim of our study was to investigate the efficacy of respiratory muscle training in children undergoing kidney transplantation.

DETAILED DESCRIPTION:
Kidney transplantation is the main treatment for patients with end-stage renal failure. Although kidney transplantation offers a good quality of life to patients, some of the complications caused by the underlying kidney disease and during end-stage renal failure persist in the follow-up of these patients, as well as many complications related to the drugs used after transplantation. As chronic kidney disease progresses, especially restrictive type respiratory dysfunction, respiratory muscle myopathy and decreased respiratory muscle strength are the most common changes seen in the pulmonary system. To improve respiratory muscle strength, respiratory muscle training is recommended for people with chronic kidney disease. There is limited scientific evidence on respiratory muscle training methods and outcomes in patients with chronic kidney disease, especially focusing only on inspiratory muscle training. Considering the heterogeneity of the studies and the variability of the results, the effectiveness of respiratory muscle training in patients with chronic kidney disease and especially after transplantation remains unclear. In the light of all this information, the aim of our study was to investigate the effectiveness of respiratory muscle training in children undergoing kidney transplantation. Patients will be randomly divided into two groups as experimental and control groups. According to the sample size calculation, it was determined that at least 15 people should be included in each group. Children in the experimental and control groups will be taught a home-based chest physiotherapy program (breathing exercises, teaching relaxation positions, cough training, respiratory control, respiratory control, physical activity recommendation) to be applied for 30 minutes a day, 5 days a week for 8 weeks. In addition to this program, patients in the experimental group will be given inspiratory and expiratory combined respiratory muscle training at 30% of MEP and MIP values for 8 weeks, 2 times a day for 20 minutes each, at least 5 days a week. The resistance setting of the patients in the experimental group will be adjusted to be calculated by measuring MIP-MEP again. Patients in the control group will receive sham combined respiratory muscle training for a total of 8 weeks at the lowest constant load, 2 times a day for 20 minutes each, at least 5 days a week.

ELIGIBILITY:
Inclusion Criteria:

* Being between 8-18 years old
* At least 6 months have passed since kidney transplantation
* Being able to walk, cooperate and clinically stable
* Volunteering to participate in the study

Exclusion Criteria:

* A history of hospitalization in the last four weeks before study participation History of hospitalization during the exercise training program
* Having secondary diseases such as kyphoscoliosis that may affect respiratory function
* Currently participating or have participated in regular exercise training in the last 1 year
* Having neurological, psychiatric, orthopedic, cardiovascular and pulmonary system comorbid conditions that prevent the performance of tests and participation in the treatment program

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Test | Eight weeks
  Change from baseline forced vital capacity (FVC) at 8 weeks.
Respiratory Function Test | Eight weeks
  Change from baseline forced forced expiratory volume in 1 (FEV1) second at 8 weeks.
Respiratory Function Test | Eight weeks
  Change from baseline peak expiratory flow (PEF) at 8 weeks.
Respiratory Function Test | Eight weeks
  Change from baseline FEV1/FVC at 8 weeks.
Respiratory Muscle Strength | Eight weeks
  Change from baseline maximum inspiratory pressure (MIP) at 8 weeks.
Respiratory Muscle Strength | Eight weeks
  Change from baseline maximum expiratory pressure (MEP) at 8 weeks.
Peripheral Muscle Strength | Eight weeks
  Change from baseline m. quadriceps strength at 8 weeks.
Peripheral Muscle Strength | Eight weeks
  Change from baseline m. biceps strength at 8 weeks.
Functional Capacity | Eight weeks
  Change from baseline distance covered in six minute walk test at 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No